CLINICAL TRIAL: NCT07080294
Title: Use of Injectable Extended Platelet-Rich Fibrin as a Local Adjunctive Therapy in the Treatment of Stage II Periodontitis Patients (Randomized Controlled Clinical Trial)
Brief Title: Use of Injectable Extended Platelet-Rich Fibrin as a Local Drug Delivery in the Treatment of Stage II Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0401024OM
Record Dates: First submitted 2025-07-13; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis Stage II; Gingival Pocket
Keywords: eprf; periodontitis stage II; Alb prf; pocket; albumin; SRP; extended prf; extended platelet rich fibrin; gel
MeSH Terms: conditions — Periodontitis; Gingival Pocket | interventions — Albumins; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- extended platelet rich fibrin injection in pocket (Experimental): Thorough periodontal mechanical debridement and injection of ePRF inside the assigned pockets will be performed for 15 patients of stage II periodontitis.
  Interventions: Other: extended platelet rich fibrin injection in pocket
- albumin injection in pocket (Experimental): Scaling and root planing and injection of albumin gel alone inside the pockets will be performed for 15 patients of stage II periodontitis
  Interventions: Other: albumin injection in pocket
- scaling and root planing (Experimental): Mechanical debridement alone will be performed for 15 patients with stage II periodontitis without injection of any material into the pockets.
  Interventions: Other: scaling and root planing

INTERVENTIONS:
Other: extended platelet rich fibrin injection in pocket — Whole blood (10 mL) will be centrifuged at 700 g for 8 minutes. The upper layer (yellow layer) shows the liquid plasma layer. The most upper layer of platelet- poor plasma (PPP) will be collected in a syringe. then PPP will be heated in a heat block device at 75°C for 10 minutes and thereafter cooled to room temperature for approximately 2 minutes. An injectable albumin gel will then be prepared. Then the liquid platelet-rich layer (liquid-PRF) including the buffy coat layer with accumulated platelets and leukocytes, will be collected in a separate syringe. The albumin gel and native liquid PRF will then be thoroughly mixed by utilizing a female-female luer lock connector. Now injectable e-PRF in final form is ready to be used.
  Arms: extended platelet rich fibrin injection in pocket
Other: albumin injection in pocket — Whole blood (10 mL) will be centrifuged at 700 g for 8 minutes. The upper layer (yellow layer) shows the liquid plasma layer. The most upper layer of platelet- poor plasma (PPP) will be collected in a syringe. then PPP will be heated in a heat block device at 75°C for 10 minutes and thereafter cooled to room temperature for approximately 2 minutes. An injectable albumin gel will then be prepared.
  Arms: albumin injection in pocket
Other: scaling and root planing — removes plaque and calculus above and below the gumline using manual or ultrasonic instruments.
  Arms: scaling and root planing

SUMMARY:
The objective of the present study is to assess the clinical effectiveness of local delivery of injectable extended platelet-rich fibrin in subgingival application when used in conjunction with scaling and root planing (SRP) in the treatment of stage II periodontitis.

The primary outcome includes the clinical attachment gain after 6 months, whereas the secondary outcomes include the changes of probing pocket depth, bleeding on probing percentage, plaque and gingival indices and the concentration of matrix metalloproteinase-8 (MMP-8) in gingival crevicular fluid (GCF) after 3 and 6 months.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory dysbiotic disease resulting in damage of the periodontal tissue surrounding the teeth. At first, the teeth loosen, and eventually, there may be tooth loss. Periodontitis occurs due to an imbalance in the oral microbiota's natural balance and host resistance (i.e., dysbiosis). In adults, dysbiosis may be the cause of periodontitis, which can lead to inflammatory changes that affect the bone and connective tissue (1, 2).

The goals of today's treatment of periodontitis are to reduce infection, resolve inflammation and create a clinical condition, which is compatible with periodontal health (3). Periodontitis is typically treated initially in a non-surgical way. Non-surgical periodontal therapy consists of scaling and root planing (SRP) combined with oral hygiene instructions. Typically, this results in clinical attachment gain due to resolution of the inflammation. However, findings revealed that in some affected areas, the standard treatment proved to be insufficient and some residual pockets remain after therapy (4).

To reduce the indication of surgical invasive and technically demanding procedures, several adjuncts to SRP have been proposed such as the use of antibiotics or anti-inflammatory drugs. These adjunctive therapies improved treatment outcomes in terms of pocket depth reduction and CAL gain (5). However, their systemic administration requires the use of high dose of active drugs to reach efficient concentration at the treated site, the compliance of the patient to follow the selected administration regimen and could be associated with serious side effects. Consequently, several local treatments such as gels, fibers or chips loaded with different active molecules or drugs have been developed and evaluated in clinical settings (6).

The main advantages of such treatments are the delivery of active drugs at the precise site of the lesions, the reduced risk of side effects and the possibility of 3D stabilization of the blood clot (7). Local application of medications after scaling and root planing (SRP) has shown better results than SRP alone principally in reduction of pocket depth (8). Nonetheless, some materials which are applied locally were found to induce allergic -like reactions, lack the rheological characteristics and sustained release of the active ingredient under investigation (9).

To-date, platelet concentrates have been proven to promote and stimulate wound healing processes and to accelerate angiogenesis due to their concentrated growth factors content and anti-inflammatory molecules. Del Fabbro and his colleagues confirmed the use of growth factors for providing an additional stimulation to physiological healing processes (10).

Platelet concentrates are classified as platelet-rich plasma (PRP) or platelet-rich fibrin (PRF). In PRP techniques, blood is collected with anticoagulant and then centrifuged, whereas in PRF techniques, blood is collected without any anticoagulant and immediately centrifuged (11).

As for leukocyte- and platelet-rich fibrin (L-PRF) products, including L-PRF clots and liquid fibrinogen, platelet concentrates are obtained by centrifugation of a whole blood sample, discarding red blood cells and concentrating the components to be used, such as fibrin, platelets, growth factors, leukocytes, and other circulating cytokines and proteins (12). Nevertheless, the common demerit of current platelet concentrates is the fast resorption within 15 days inside the site of application (13).

Recently, a new PRF preparation has been introduced by Richard Miron (2020) known as extended platelet- rich fibrin (e-PRF) or Albumin-PRF mixture (Alb-PRF). It consists of a combination of concentrated growth factors and denaturated albumin gel. It is postulated that it might resorb after 4-6 months; therefore, it can be used even for guided bone regeneration (14) .

Extended platelet- rich fibrin (ePRF) is the latest functional and promising matrix that overcomes limitations of its predecessors. It shows many characteristics of ideal biomaterial for repair, regeneration, or facial esthetics. Here are some important characteristics: it is injectable which allows physicians to minimize access trauma to affected tissue and there is no need for sophisticated armamentarium for its production as a chairside procedure in the clinics (15).

ePRF can be used as a bioactive, natural filler as it forms a "sticky" gel that can be used as a 100% natural filler and it does not easily leak out from the injury site. Its gel creates a natural scaffold allowing absorption of water that is necessary for proliferation of new cells. It does not block the space for newly formed tissue (16).

Thus, the alternative hypothesis of the present study states that the injectable extended platelet rich fibrin could improve the periodontal status of patients who are suffering from stage II periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage II Periodontitis (pocket depth ≤ 5mm and CAL = 3-4 mm).
2. Age range (30-50) years.
3. Good compliance with the plaque control instructions following initial therapy.
4. Availability for follow- up and maintenance program.

Exclusion Criteria:

1. Periodontitis patients with stage I, III and IV.
2. Smoking.
3. Systemic diseases which could influence the outcome of the therapy.
4. Pregnant and lactating females.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
clinical attachment gain | 6 months
  Clinical Attachment Level (CAL) measured from the cementoenamel junction to the base of the gingival sulcus (RD+PD).

SECONDARY OUTCOMES:
Probing Depth (PD) | 6 months
  The assessment of probing pocket depth involved measuring the distance from the free gingival margin to the base of the pocket using a 1 mm UNC 15 periodontal probe, which was inserted into the gingival sulcus parallel to the tooth's long axis. Readings were documented from three buccal sites-mesiobuccal, middle-buccal, and distobuccal-and three lingual sites-mesial-lingual, middle-lingual, and distal-lingual. The probing depths recorded (3-5 mm) were summed and divided by the total number of pockets to derive the mean probing pocket depth for each patient.
Plaque index (PI). | 6 months
  According to the Silness and Loe plaque index (1964), the cervical plaque level was determined by measuring soft deposit thickness, excluding coronal plaque extension. The scoring process utilized a UNC 15 periodontal probe (1 mm), dental mirrors, sharp explorers, and appropriate lighting, with an air jet applied to dry teeth and gingival tissues before evaluation.
Gingival index | 6 months
  The Löe and Silness index (1963) serves as a tool for examining gingival conditions by tracking qualitative changes. It evaluates the severity and spread of gingivitis, focusing on four designated sites per tooth, including the distofacial and mesiofacial papillae, the facial gingival margin, and the lingual gingival margin
Bleeding on probing (BOP) | 6 months
  A follow-up evaluation, the study further investigates bleeding on probing (BOP) as a clinical determinant of either periodontal disease progression or stability. The presence or absence of BOP is a well-established criterion for diagnosing periodontal health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, DK, Egypt